CLINICAL TRIAL: NCT06692712
Title: Intrathecal Administration of MELPIDA (AAV9/AP4M1) For Hereditary Spastic Paraplegia Type 50 (SPG50): A Phase 3, Open-Label Trial With Matched Prospective Concurrent Control Arm
Brief Title: Phase 3 Efficacy Study With Concurrent Control of IT MELPIDA in SPG50.Concurrent Controls.
Acronym: SPG50
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Elpida Therapeutics SPC (Industry)
Collaborators: University of Texas Southwestern Medical Center (Other); Hospital Sant Joan de Deu (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MELPIDA -Pivotal Trial
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Hereditary Spastic Paraplegia Type 50
Keywords: SPG50; Spastic Paraplegia; Gene Therapy; Phase 3
MeSH Terms: conditions — Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MELPIDA Treatment (Experimental): Eligible subjects (N=8) will receive a single open-label intrathecal administration of MELPIDA and follow up to week 260.
  Interventions: Genetic: MELPIDA
- Matched Prospective Concurrent Control Arm (No Intervention): Approximately 16 untreated age- and disease- matched controls with confirmed AP-4-related disease (SPG47, SPG50, or SPG52) will be enrolled and attend study visits concurrent with the MELPIDA treatment arm.

INTERVENTIONS:
Genetic: MELPIDA — Gene Therapy agent
  Arms: MELPIDA Treatment

SUMMARY:
Phase 3, open-label study to assess the efficacy and safety of a single lumbar intrathecal administration of MELPIDA in individuals with Hereditary Spastic Paraplegia Type 50 (SPG50).

DETAILED DESCRIPTION:
MELPIDA is an AAV9-based gene therapy vector that expresses the fully functional form of AP4M1 under the control of a synthetic promoter. MELPIDA will be delivered intrathecally and is designed to achieve stable, potentially life-long expression of AP4M1 in non-dividing cells. This clinical study is a pivotal open-label phase 3 study designed to assess safety and efficacy of MELPIDA in individuals with SPG50.

ELIGIBILITY:
To be eligible to participate in this study candidates must meet the following eligibility criteria at Screening:

Inclusion:

For the treatment group

* Male and females between the ages of 4 months to 72 months at the time of screening.
* Molecularly-confirmed diagnosis of SPG50 (confirmed by a CLIA certified, CE-marked, or equivalent lab): Genomic DNA mutation analysis demonstrating bi-allelic pathogenic variants in the AP4M1 gene.
* Subjects must have features of neurologic dysfunction by clinical history and physical examination.
* Stable doses of concomitant medications such as anti-spasticity medications, anti-seizure medications, behavioral management medications, sleep medications, and special diets, supplements, or nutritional support for at least 3 months prior to Screening. If recent changes (< 3 months) in medications, the subject may be allowed per Investigator judgement.
* Parent/legal guardian willing to provide written informed consent for their child prior to participation in the study,
* Subjects and caregivers must demonstrate ability to travel to the study center. For the 30 days post treatment subjects must reside within 100 miles (approximately 160 km) of the clinical site.

For the control group

* Male and females between the ages of 4 to 72 months at the time of screening.
* A molecularly confirmed diagnosis of SPG47, SPG50 or SPG52 (confirmed by a CLIA certified, CE-marked, or equivalent lab). Genomic DNA mutation analysis demonstrating bi-allelic pathogenic variants in the AP4B1, AP4M1, or AP4S1 gene,
* Subjects must have features of neurologic dysfunction by clinical history and physical examination.
* Parent/legal guardian willing to provide written informed consent for their child prior to participation in the study.
* Subject able to comply with all protocol requirements and procedures.
* Subjects and caregivers must demonstrate the ability to travel to the study center.

Exclusion:

For the treatment group

* Inability to participate in the clinical evaluation as determined by the principal investigators.
* Clinically significant abnormal laboratory values (hemoglobin < 6 or > 20 g/dL; white blood cell > 20,000 per cmm, platelets count < 100,000 per cmm; INR > ULN; GGT, ALT, and AST or total bilirubin > 1.5 × ULN, creatinine ≥ 1.5 mg/dL) prior to gene replacement therapy.
* Presence of a concomitant medical condition (eg, scoliosis or bleeding disorder) that precludes a lumbar puncture or use of anesthetics for sedated procedures.
* Documented cardiomyopathy or significant congenital heart abnormalities.
* History of severe/life-threatening allergic reaction to sirolimus, tacrolimus, corticosteroids, or gadolinium.
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer, or interactions with the immunosuppressive agents.
* Any item which would exclude the subject from being able to undergo MRI according to local institutional policy, or any other procedure.
* The presence of significant AP-4 related CNS impairment or behavioral disturbances that would confound the scientific rigor or interpretation of results of the study.
* Recent or planned elective surgical procedures (within 6 months) that would confound the scientific rigor or interpretation of results of the study.
* Failure to obtain appropriate informed consent.
* Reason to believe that the subject or parents of the subject will not comply with the study procedures outlined in the study protocol.
* Have received an investigational drug within 30 days prior to screening or plan to receive an investigational drug (other than gene therapy) during the study.
* Enrollment and participation in another interventional clinical trial 90 days before first visit (screening).

For the control group

* Inability to participate in the clinical evaluation as determined by the principal investigators.
* Any other situation that would exclude the subject from undergoing any other procedure required in this study.
* The presence of significant AP-4 related CNS impairment or behavioral disturbances that would confound the scientific rigor or interpretation of results of the study.
* Recent or planned elective surgical procedures that would confound the scientific rigor or interpretation of results of the study.
* Failure to obtain appropriate informed consent.
* Reason to believe that the subject or parents of the subject will not comply with the study procedures outlined in the study protocol.
* Have received an investigational drug within 30 days prior to screening or plans to receive an investigational drug (other than gene therapy) during the study.
* Enrollment and participation in another interventional clinical trial 90 days before first visit (screening).

Ages: 21 Months to 78 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2032-02-28 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-88) Defined Major Milestones | 156 weeks
  Change in total percent score of the 8 Major Motor Milestone Scores from baseline in treated group compared to change in total percent score of the 8 Major Motor Milestone Scores from baseline in untreated controls
  1. #24: Sit on mat: Maintain, arms free, 3 seconds
  2. #38: Prone: Creeps forward 1.8m (6')
  3. #52: On the floor: Pulls to stand at large bench
  4. #67: Standing: 2 hands held: walks forward 10 steps
  5. #69: Standing: Walks forward 10 steps
  6. #84: Standing: Holding 1 rail: walks up 4 steps, holding 1 rail, alternating feet
  7. #85: Standing: Holding 1 rail: walks down 4 steps, holding 1 rail, alternating feet
  8. #88: Standing on 15cm (6") step: Jumps off, both feet simultaneously

SECONDARY OUTCOMES:
Composite Endpoint Defined by the Win Ratio | 156 weeks
  Composite Endpoint Defined by the Win Ratio using matching criteria after 156 Weeks of Follow-up of the 8 selected items and the raw scores of the Cognitive domain of the Bayley Scale of Infant and Toddler Development 4th Edition (Bayley-4).
Developmental Milestones- Bayley-4 Cognitive Domain | 156 weeks
  Developmental Milestones- Bayley-4 Cognitive Domain-Change in Total Raw Score from Baseline
Gross and Fine Motor Function (GMFM-88 full scale) | 156 weeks
  Gross and Fine Motor Function (GMFM-88 full scale) - Change in Total Score from Baseline.
Disease Severity (Spastic Paraplegia Rating Scale ) | 156 weeks
  Disease Severity (Spastic Paraplegia Rating Scale ). Change in Total Score from Baseline.
Disease Severity (Clinical Global Impression) | 156 weeks
  Disease Severity (Clinical Global Impression) Change in Physician-assessed Clinical Global Impression) from Baseline.
Muscle Spasticity (Modified Ashworth Scale) | 156 weeks
  Change from Baseline in Muscle Spasticity (Modified Ashworth Scale) Score

CONTACTS AND LOCATIONS:
Locations (2):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States
- Sant Joan de Deu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Will be posted on Elpida Therapeutics website
Supporting Information: Study Protocol, CSR
Time Frame: 12 months after start date for protocol. CSR 12 months after completion of study

REFERENCES:
- [Derived] Agianda HAP, Kim HM, Battaglia N, Rong J, Tam A, Gonzalez Saez-Diez E, Boerkoel CF, Saffari A, Quiroz V, Schierbaum L, Zaman Z, Bernardi K, Ebrahimi-Fakhari D. Diagnostic Utility of the ATG9A Ratio in AP-4-Associated Hereditary Spastic Paraplegia. Ann Clin Transl Neurol. 2026 Jan 5. doi: 10.1002/acn3.70308. Online ahead of print. PMID 41491634